CLINICAL TRIAL: NCT00841048
Title: A Randomised, Single-blind, Placebo-controlled, Single Centre, Phase I Study in Healthy Volunteers to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD4017 After Repeated Ascending Oral Doses
Brief Title: Phase I Study in Healthy Volunteers to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD4017 After Repeated Ascending Oral Doses
Acronym: MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Jan Eriksson MD PhD / Medical Science Director, AstraZeneca R&D Mölndal, Sweden
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: D2060C00002
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Safety and tolerability
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 2-(1-(5-(cyclohexylcarbamoyl)-6-propylsulfanylpyridin-2-yl)-3-piperidyl)acetic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD4017 in ascending doses (start dose 75mg od)
  Interventions: Drug: AZD4017
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD4017 — ascending multiple doses(start dose 75mg od), oral suspension
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The primary aim of this study is to investigate the safety and tolerability of AZD4017 when given as multiple oral ascending doses to healthy volunteers. This will be done by comparing the effect of AZD4017 to placebo. The study will aslo investigate the absorption, distribution and disappearance of AZD4017 in the body. Information about plasma concentrations of AZD4017 vs time after dose intake will also be collected and some measures of pharmacokinetics versus pharmacodynamics will be included. The future indication for AZD4017 is planned to be Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written and dated informed consent
* BMI between 19 and 30 kg/m2
* Subjects must be willing to use barrier methods of contraception

Exclusion Criteria:

* History of any clinically significant disease
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of investigational product
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Laboratory blood sample result showing elevated liver enzymes (ASAT, ALAT) and muscle enzymes (CK).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2009-02; Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability (Adverse events, vital signs, ECGs, physical examination, laboratory variables | The variables will be measured predose and then repeatedly during the study

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax), time to Cmax (tmax), terminal half-life, area under the plasma concentration-time curve and the apparent oral plasma clearance (CL/F) | Blood samples for determination of AZD4017 concentration will be taken predose and repeatedly during the study.
Laboratory screen to evaluate effect on metabolic variables | Blood samples will be taken pre-dose and repeatedly during the study
Pharmacodynamic measurements allowing to assess AZD4017 effect in different tissues | Baseline and repeatedly after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Hartford, MD PhD, Principal Investigator — AstraZeneca Clinical Pharmacolgy Unit Sahlgrenska University Hospital SE-413 45 Göteborg Sweden
Locations (1):
- Research Site, Gothenburg, Sweden